CLINICAL TRIAL: NCT01119183
Title: Improving Patient Understanding of Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00006039
Record Dates: First submitted 2010-04-23; First posted 2010-05-07 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Preeclampsia
Keywords: Patient understanding and counseling
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention)
- 2 (Active Comparator)
  Interventions: Behavioral: ACOG education pamphlet on preeclampsia
- 3 (Experimental)
  Interventions: Behavioral: Preeclampsia education tool

INTERVENTIONS:
Behavioral: ACOG education pamphlet on preeclampsia — The ACOG pamphlet on preeclampsia will be offered to this group
  Arms: 2
Behavioral: Preeclampsia education tool — The newly created preeclampsia educational tool will be offered to this group
  Arms: 3

SUMMARY:
Participants counseled with the preeclampsia educational tool will have a better understanding of preeclampsia than those not counseled using the tool.

ELIGIBILITY:
Inclusion Criteria:

* 12-40 weeks pregnant
* No significant hearing or vision impairment
* English speaking

Exclusion Criteria:

* Active diagnosis of preeclampsia
* Significant hearing or vision impairment
* Non-English speaking

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Improved understanding of preeclampsia | one week
  Understanding of preeclampsia will be assessed through a questionnaire that asks a series of closed ended questions about preeclampsia as well as a single open ended question. This questionnaire has been used in a prior study and has proven to be a useful assessment of patient knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] You WB, Wolf MS, Bailey SC, Grobman WA. Improving patient understanding of preeclampsia: a randomized controlled trial. Am J Obstet Gynecol. 2012 May;206(5):431.e1-5. doi: 10.1016/j.ajog.2012.03.006. Epub 2012 Mar 13. PMID 22542120